CLINICAL TRIAL: NCT04225234
Title: Sustaining the Reach of a Scalable Weight Loss Intervention Through Financial Incentives: an Exploratory Randomized Controlled Trial
Brief Title: Sustaining the Reach of a Scalable Weight Loss Intervention Through Financial Incentives
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the COVID-19 pandemic
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0211-19-EP
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Overweight and Obesity
Keywords: Financial incentive; Behavioral economics; Attrition; Reach; Participation; Retention; Weight loss
MeSH Terms: conditions — Overweight; Obesity; Tooth Wear; Weight Loss

STUDY DESIGN:
Intervention Model Description: Our proposed project would be most appropriately be categorized as a partial factorial with choice model, because our study design includes 2 intervention each alone (weight loss and weigh-in), and in combination (weight loss + weigh-in), and choice. No control group is included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Weight loss incentive (Active Comparator): Participants will receive incentive rewards based on WEIGHT LOSS outcomes.
  Interventions: Other: Financial incentives
- Weigh-in incentive (Experimental): Participants will receive incentive rewards based on WEIGH-INs frequency
  Interventions: Other: Financial incentives
- Combination incentive (Experimental): Participants will receive half of the incentive from WEIGHT LOSS and WEIGH-INs
  Interventions: Other: Financial incentives
- Choice option incentive (Experimental): Participants will choose one out of the three incentive programs (Weight-loss, Weigh-ins, and Combination).
  Interventions: Other: Financial incentives

INTERVENTIONS:
Other: Financial incentives — Depending on their level of participation or weight loss outcomes, participants will have the opportunity to receive between $60-$120 (over 12 months), on average, regardless of program assignment.
  Regardless of which incentive program that participants are randomized to, they will receive the incentaHEALTH weight loss program intervention. incentaHEALTH is an technology-supported multi-component coaching intervention for weight loss includes a website, objective weight assessment using HIPAA-compliant kiosks, daily social cognitive theory-based email and text message support, and online access to health coaches. The intervention encourages increased intake of fruit, vegetables, lean protein, and complex carbohydrates while monitoring portion sizes.

SUMMARY:
This study seeks to assess how different incentive strategies may reduce the initial attrition gap when implementing weight management in a primary care clinic predominantly serving African American patients. This will be done through an innovative research-practice partnership involving primary care, research expertise, and a small business. Participants will be randomly assigned to one of four financial incentive conditions respectively tied to: weight loss, weigh-ins, weigh-ins and weight-loss, and incentive choice. Participants will be followed for 3 and 6 months to assess program reach, sustaining the reach after initial weigh-in, and weight loss outcomes based on records on participant enrollment and subsequent weigh-ins automatically collected through a kiosk at the clinic.

DETAILED DESCRIPTION:
The proposed study "Sustaining the Reach of a Scalable Weight Loss Intervention through Financial Incentives: an Exploratory Randomized Trial" seeks to assess how the use of different incentive strategies may reduce the initial attrition gap when implementing weight management in a primary care clinic predominantly serving African American patients through an innovative research-practice partnership involving primary care, research expertise, and a small business.

The sample will include approximately 200 persons ages 19+ from Nebraska Medicine or the greater Omaha community. The inclusion criteria are (1) age 19+ years; (2) are obese (BMI >=30) or overweight (BMI >=25 yet smaller than 30); (3) have internet access. Following the completion of an automated informed consent embedded within the program registration using a kiosk placed at the Fontenelle Clinic, we plan to conduct a 4-arm, pragmatic randomized controlled trial (RCT) that will randomly assign overweight/obese patients at the Nebraska Medicine Fontenelle clinic to one of four financial incentive conditions respectively tied to: weight loss, weigh-ins, weigh-ins and weight-loss, and incentive choice, following the completion of an automated informed consent embedded within the program registration and initial weigh-in. Participants will be followed for 3 and 6 months to assess program reach, sustaining the reach after initial weigh-in, and weight loss outcomes based on records on participant enrollment and subsequent weigh-ins automatically collected through a kiosk placed at the Fontenelle clinic.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese participants who are of 19 years or older and have internet access

Exclusion Criteria:

* Not meeting the inclusion criteria.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Sustaining the reach | 3, 6, and 12 months
  Percentage of participants returning to weigh-in 3, 6, and 12 months after initial program registration

SECONDARY OUTCOMES:
Weight loss | 3, 6, and 12 months
  weight loss achieved at 3, 6 and 12 months
Clinical meaningful weight loss | 3, 6, and 12 months
  Percentage of participants achieving clinically significant weight loss (percentage of patients who lost >3% or >5% of their initial bodyweight)

CONTACTS AND LOCATIONS:
Overall Officials: Tzeyu Michaud, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Nebraska Medicine Fontenelle clinic, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Michaud TL, Estabrooks PA, You W, McGuire TJ, Almeida F, Karls K, Love K, King K, Hill J, Reed J, Porter G, Su D. Sustaining the reach of a scalable weight loss intervention through financial incentives- a pragmatic, feasibility, online randomized trial protocol. Contemp Clin Trials. 2020 Nov;98:106142. doi: 10.1016/j.cct.2020.106142. Epub 2020 Sep 10. PMID 32920241